CLINICAL TRIAL: NCT01014754
Title: Nephrogenic Systemic Fibrosis and Gadolinium-A Medical Record Review With Analysis of Existing Skin and Other Tissue Specimens to Assess Potential Causative or Associated Factors
Brief Title: Nephrogenic Systemic Fibrosis (NSF): Analysis of Tissue Gadolinium Levels
Acronym: NSF
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Anne Laumann, Professor of Dermatology, Northwestern University
Other Study IDs: STU1460; NIH Grant #2 R01 CA102713-03A2
Record Dates: First submitted 2009-11-13; First posted 2009-11-17 (Estimated); Last update posted 2014-12-04 (Estimated); Status verified 2014-12

CONDITIONS: Nephrogenic Systemic Fibrosis; Nephrogenic Fibrosing Dermopathy
MeSH Terms: conditions — Nephrogenic Fibrosing Dermopathy

STUDY DESIGN:
Observational Model: Case-Control
Biospecimen Retention: Samples With DNA — Existing skin tissue from standard of care biopsies
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (6):
- NSF: Biopsy-proven diagnosis of NSF
- Kidney dysfunction plus gadolinium exposure: Those on dialysis or with eGFR ≤ 30 ml/min/1.73 m2 who have had a medical imaging procedure using GBCA in the 2 years prior to skin biopsy.
- Kidney dysfunction without gadolinium exposure: Those on dialysis or with eGFR ≤ 30 ml/min/1.73 m2 who have never been exposed to GBCA and have had skin biopsy.
- Normal kidney function with gadolinium exposure: Those with normal kidney function who have undergone a medical imaging procedure using Gd-based contrast agent (GBCA) in the 2 years prior to a skin biopsy.
- Normal kidneys without gadolinium exposure: Those with normal kidney function who have never been exposed to GBCA and have had a skin biopsy.
- Controls: Existing skin tissue from neonatal skin (<6 months) will be used as controls, as they presumably have never been exposed to gadolinium

SUMMARY:
The primary objective of this study is to determine any causative or associated factors for the development of Nephrogenic Systemic Fibrosis (NSF), Nephrogenic Fibrosing Dermopathy (NFD), or related diagnosis. Our primary focus will be on the previous administration of gadolinium to these patients, but we will also look at other postulated causes and risk factors.

The secondary objective of this study is to assess tissue gadolinium (Gd) levels in five groups of subjects:

* Those affected by NSF.
* Those with normal kidney function who have undergone a medical imaging procedure using Gd-based contrast agent (GBCA) in the 2 years prior to a skin biopsy.
* Those with normal kidney function who have never been exposed to GBCA and have had a skin biopsy.
* Those on dialysis or with eGFR ≤ 30 ml/min/1.73 m2 who have had a medical imaging procedure using GBCA in the 2 years prior to skin biopsy.
* Those on dialysis or with eGFR ≤ 30 ml/min/1.73 m2 who have never been exposed to GBCA and have had skin biopsy.

We hypothesize that there is a correlation between the administration of Gd-containing agents usually associated with MRI procedures and the development of NSF in those with renal failure and some other predisposing condition. We also hypothesize that tissue Gd levels in those with NSF will be higher than in those who have been exposed to GBCA but do not have NSF. Of the two groups without NSF but with exposure to GBCA, we hypothesize that those with kidney dysfunction will have higher tissue Gd levels than those with normal kidney function. We hypothesize that in the two groups of subjects without exposure to GBCA, there will be no detectable levels of Gd, regardless of kidney function status.

ELIGIBILITY:
NSF group

Inclusion Criteria:

* Biopsy-confirmed diagnosis of NSF

Exclusion Criteria:

* Does not have NSF

Normal renal plus gadolinium exposure

Inclusion Criteria:

* eGFR >30
* Existing skin tissue sample
* Gadolinium exposure in 2 years preceding skin biopsy

Exclusion Criteria:

* Does not fit inclusion criteria

Abnormal renal plus gadolinium exposure

Inclusion Criteria:

* eGFR <30 or on dialysis
* Existing skin tissue sample
* Gadolinium exposure in 2 years preceding skin biopsy

Exclusion Criteria:

* Does not fit inclusion criteria

Abnormal renal without gadolinium exposure

Inclusion Criteria:

* eGFR <30 or on dialysis
* Existing skin tissue sample
* No gadolinium exposure ever

Exclusion Criteria:

* Does not fit inclusion criteria

Normal renal without gadolinium exposure

Inclusion Criteria:

* eGFR >30
* Existing skin tissue sample
* No gadolinium exposure ever

Exclusion Criteria:

* Does not fit inclusion criteria

Controls (neonatal)

Inclusion Criteria:

* Existing skin biopsy tissue that was performed within the first 6 months of life

Exclusion criteria:

* Does not fit inclusion criteria

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Those with NSF (25). 40 subjects selected through Northwestern University Department of Dermatology's existing medical records and pathology specimens. Medical records will be reviewed to identify 10 subjects who have had a standard of care skin biopsy in the dermatology clinics at Northwestern University and who were exposed to Gadolinium in the 2 years prior to skin biopsy. Another 10 subjects who have had skin biopsy and who have never been exposed to GBCA during a medical imaging procedure will also be identified. Another 10 subjects on dialysis or with eGFR ≤30 exposed to GBCA in the 2 years prior to skin biopsy will be identified. Another group of 10 subjects on dialysis or with eGFR ≤30 who have had skin biopsy and who have never been exposed to GBCA during a medical imaging procedure will also be identified. Neonatal skin tissue of up to 10 subjects with existing skin tissue sample will be sent for analysis.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2007-08; Primary Completion 2014-04 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
To determine causative or associated factors for the development of Nephrogenic Systemic Fibrosis (NSF), Nephrogenic Fibrosing Dermopathy (NFD), or related diagnosis. | 1988 to present

SECONDARY OUTCOMES:
Tissue Gadolinium Level in 5 groups of patients, with and without NSF | 1988 to present
  * Those affected by NSF.
  * Those with normal kidney function who have undergone a medical imaging procedure using Gd-based contrast agent (GBCA) in the 2 years prior to a skin biopsy.
  * Those with normal kidney function who have never been exposed to GBCA and have had a skin biopsy.
  * Those on dialysis or with eGFR ≤ 30 ml/min/1.73 m2 who have had a medical imaging procedure using GBCA in the 2 years prior to skin biopsy.
  * Those on dialysis or with eGFR ≤ 30 ml/min/1.73 m2 who have never been exposed to GBCA and have had skin biopsy.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Laumann, MBChB, MRCP(UK), Principal Investigator — Northwestern University
Locations (1):
- Northwestern University Feinberg School of Medicine, Department of Dermatology, Chicago, Illinois, United States

REFERENCES:
- [Background] High WA, Ayers RA, Chandler J, Zito G, Cowper SE. Gadolinium is detectable within the tissue of patients with nephrogenic systemic fibrosis. J Am Acad Dermatol. 2007 Jan;56(1):21-6. doi: 10.1016/j.jaad.2006.10.047. Epub 2006 Nov 9. PMID 17097388
- [Background] Khurana A, Greene JF Jr, High WA. Quantification of gadolinium in nephrogenic systemic fibrosis: re-examination of a reported cohort with analysis of clinical factors. J Am Acad Dermatol. 2008 Aug;59(2):218-24. doi: 10.1016/j.jaad.2008.04.010. Epub 2008 Jun 5. PMID 18538448
- [Background] Cowper SE, Robin HS, Steinberg SM, Su LD, Gupta S, LeBoit PE. Scleromyxoedema-like cutaneous diseases in renal-dialysis patients. Lancet. 2000 Sep 16;356(9234):1000-1. doi: 10.1016/S0140-6736(00)02694-5. PMID 11041404